CLINICAL TRIAL: NCT05209178
Title: Diagnostic Accuracy of Self-collected Versus Healthcare Collected Anterior Nose Swabs for SARS-CoV-2 Detection - a Randomized Controlled Trial.
Brief Title: Diagnostic Accuracy of Self-sampling Versus Healthcare Sampling for Coronavirus-Disease-2019 Detection.
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Emergency Medical Services, Capital Region, Denmark (Other Government); Technical University of Denmark (Other); Copenhagen Medical A/S (Unknown)
Responsible Party: Principal Investigator, Kathrine Kronberg Jakobsen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CVB2022 - CoV2 selftest
Record Dates: First submitted 2022-01-14; First posted 2022-01-26 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 Serological Testing; Rapid Antigen Test; Self-collected specimen
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-collection of specimen (Experimental): Participants allocated to this arm will perform specimen collection for the antigen tests independently using written instructions and access to a video. Sampling is performed as two individual procedures from the anterior part of the nose and the oropharynx respectively.
  Interventions: Diagnostic Test: Collection of nasal and oropharyngeal specimen for COVID19 antigen test
- Healthcare-collection of specimen (Active Comparator): Participants allocated to this arm will initially have specimen collection for the antigen tests done by a healthcare personnel. Sampling is performed as two individual procedures from the anterior part of the nose and the oropharynx respectively.
  Interventions: Diagnostic Test: Collection of nasal and oropharyngeal specimen for COVID19 antigen test

INTERVENTIONS:
Diagnostic Test: Collection of nasal and oropharyngeal specimen for COVID19 antigen test — Regarding two independent sampling procedures from the anterior part of the nose and the oropharynx, participants are randomized to either perform the sampling by themselves with written instructions or having the procedure performed by trained personnel. The specimen is meant for a rapid antigen test for COVID-19 infection.
  Other Names: Standard Q COVID-19 Ag-test, SD Biosensor INC

SUMMARY:
The current Coronavirus Disease 2019 (COVID-19) pandemic continues to be a worldwide health emergency. To contain the spread of disease, high demands on testing availability and capacity are observed. Although polymerase chain reaction (PRC) is the golden standard method in detecting infection with COVID-19, the procedure is time consuming and requires healthcare personnel and laboratories. Rapid antigen tests, however, have several potential benefits including greater scalability and results are provided much quicker. So far, sampling for rapid antigen tests is predominantly performed by health care personnel. Though, the testing and analyzing procedure of an antigen test seems manageable by laymen but the validity of a self-performed rapid antigen test is sparsely examined. Thus, the investigators wish to conduct a study evaluating the diagnostic accuracy of self-performed rapid antigen test for detecting COVID-19 infection by comparing self-performed and healthcare-performed rapid antigen tests on the same individual while using a PCR tests as a control.

DETAILED DESCRIPTION:
Background:

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the resulting COVID-19 pandemic continue to be a worldwide health emergency resulting in national lockdown.

A strategy for the opening of society has been proposed to be extensive testing.

The golden standard for correct detection of SARS-CoV-2 is by reverse transcriptase polymerase chain reaction (RT-PCR) of an upper respiratory specimen. However, this requires laboratory facilities and the test is time-consuming. Rapid antigen tests offer a simpler approach, and test results are available within minutes. Especially the latter can potentially lead to a faster containment of infection in the society. So far, the specimens for the rapid antigen test have primarily been collected by nasopharyngeal swabs by trained personnel.

Self-collected swab offers a possibility to increase testing access and would enable testing outside the healthcare system. Furthermore, self-collected swabs could lower the exposure risk of healthcare workers and could reduce the expenses for personal protective equipment, and lastly self-collection is furthermore reported as the preferred sampling method. However, self-collected swabs may pose issues of increased risk of incorrect sampling as sampling is unsupervised and the sensitivity of the self-collected tests compared to professional-collected tests has been questioned due to varying results. Studies on the rapid antigen test and self-collected swabs as a screening tool are sparse.

The aim of the study is to compare the diagnostic accuracy of self-testing for SARS-CoV-2 to a test performed by trained personnel. Both the self-collected and the collection by trained personnel will be two independent SARS-CoV-2 rapid antigen tests (Standard Q COVID-19 Ag - test, SD Biosensor INC.) by sampling from both the anterior part of the nose as well as the oropharynx. The diagnostic accuracy of the two antigen tests will furthermore be compared to a RT-PCR test based on a swab from the oropharynx.

Method

Study design:

The project is a comparative, prospective, randomized, diagnostic accuracy study.

Participants:

Citizens who have booked an appointment and show up for a COVID-19 test at Test Center, Valby, in the Capital Region are offered to participate in the project on a volunteer basis.

In Denmark, citizens are tested for infection with SARS-CoV-2 by swabs in the oropharynx, and subsequent analysis of the specimens by a RT-PCR test. The results of the swabs are given within 48 hours. The sampling procedure is performed by trained personnel. The oropharyngeal swab is a swab of the palatine tonsils and the posterior wall of the pharynx examined by RT-PCR for SARS-CoV-2.

Interventions:

Participants will, in addition to the oropharyngeal swab they are already scheduled for, be examined by swabs from the anterior part of the nose, both performed by self-collection and by a trained personnel. Participants are randomized in a 1:1 ratio between the order of the collection method from the sampling from the anterior part of the nose, respectively self-collection and collection by trained personnel.

The swabs from the anterior part of the nose and the oropharynx are analyzed by a rapid antigen test (Standard Q COVID-19 Ag - test, produced by SD Biosensor INC.). The swab of the anterior part of the nose is inserted approximately 1 inch/2 cms or until resistance in both nostrils with the same swab and are examined immediately after collection according to the manufacturer's instructions. Oropharyngeal sampling is performed by collecting specimen from the posterior wall of the oropharynx and both tonsils using a swab. This sample is analyzed alike the rapid antigen test from the anterior part of the nose. Participants are instructed in the self-sampling by means of written instructions and have the opportunity to see a tutorial video accessed by a QR-code.

The results of the swabs will be available within 15 minutes and participants will be able to see the results electronically.

The participants are registered by the Region's test staff in a secure web database (REDCap) on-site and are asked to fill out an online survey regarding information on their symptoms and vaccination status.

The leftover material of the antigen tests is afterward placed in separate tubes with virus inactivating preservation transport media. SAll samples meant for RT-PCR analysis are sent to the test facility at the Technical University of Denmark (DTU) for SARS-CoV-2 RT-PCR testing targeting two segments of the Nuceloprotein gene. Analysis results are electronically transferred to Department of Clinical Microbiology at Rigshospitalet that is responsible for the interpretation and reporting of the final result to the participant.

Clinical outcome:

The investigators will define a participant with an RT-PCR positive result as having a COVID-19 infection and this will be the diagnostic reference standard to calculate the accuracy for the self-collected rapid antigen test. The criteria for a positive RT-PCR test result will be a cycle threshold (Ct) value below 34 for at least one gene-targets for SARS-CoV2. .

Sample size:

Based on previous studies the investigators expect that the sampling performed by trained personnel have a 5% higher sensitivity than self-sampling. The investigators estimate that a sample of 1225 participants would provide the trial with an 80% power at a 5% significance level. The investigators thus wish to include a total of 8000 participants. The prevalence of COVID-19 in Denmark is currently approximately 9.3%, thus the investigators expect to have approximately 700 COVID-19 positive patients.

Randomization sequence:

The randomization is generated by a computer program (https://www.sealedenvelope.com/simple-randomiser/v1/lists). Participants are randomized at enrollment in block sizes of 40 participants. This table with randomization numbers is only available to specified personnel at the Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet.

Statistics:

The investigators wish to calculate the sensitivity and specificity with 95% confidence interval of the self-collected rapid antigen test with reference to a rapid antigen test collected by healthcare. The rate of SARS-CoV-2 detection by the two rapid antigen test collection methods will be compared using McNemar's test. The level of statistical significance is p < 0.05.

The research group:

The research group at the Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet, led by professor, Christian von Buchwald, MD., has already substantial experience in COVID-19 research, including a well-discussed study regarding the effectiveness of facial masks and a study on sensitivity of self-collective swabs, in addition to ongoing projects on impaired sense of smell and COVID-19 infection among hospital staff. The research group has recently performed a large study on the sensitivity and specificity of the rapid antigen test with swabs collected in the nasopharynx. This project will be a collaboration with a private provider, Copenhagen Emergency Medical Services. The private provider in Denmark of SD Biosensor INC., Copenhagen Medical, will provide rapid antigen tests for the collection of the rapid antigen tests.

Practical aspects of the project:

Testcenter Danmark will provide the staff required for collecting swabs for RT-PCR tests at their test sites in the Capital Region and will deliver the results from here.

In addition, an agreement has been made with Copenhagen Medical who will deliver the rapid antigen test (Standard Q COVID-19 Ag - test, produced by SD Biosensor INC.) to the test centers where the project is carried out.

Ethical considerations:

The project will provide essential knowledge regarding the sensitivity and specificity of the possibility of self-testing for COVID-19 by rapid antigen test, as an alternative to healthcare collected tests, during the current pandemic in Europe. If the sensitivity of the quick tests is high, and a more widely use is implemented, it can potentially lead to a faster containment of the COVID-19 infection in the society.

Participation in the project might be associated with a small amount of discomfort due to the collection of specimens, but no greater discomfort than otherwise associated with swabs for COVID-19. As the patients already have booked an appointment for COVID-19 testing it is expected that participants will agree with this and the investigators are thus expecting a high participation rate. There are no known risks associated with participation in the project.

The protocol complies with the Declaration of Helsinki II. Furthermore, the project is approved by the Scientific Ethics Committee.

Recruitment of participants and informed consent:

All patients older at the age of 16 years or older, who have booked an appointment for COVID-19 test, at Testcenter Danmark's test centers in the Capital Region are offered to participate in the project.

The participants will receive oral and written information about the project, as well as written information about subjects' rights. The right to bring a counsel to the information interview will likewise be explained.

The information interview is carried out by the staff from the Capital Region. Patients are offered 24 hours reflection time if needed before written consent is obtained. The participants are informed that they can withdraw their consent at any time without the affection of further processes or potential treatment.

Patients' physical and mental integrity as well as privacy:

Each participant is required to give written informed consent before he/she can be included in the study. Information obtained about participants' health, other purely private matters, and other confidential information is covered by professional secrecy.

Furthermore, patients are covered by the Health Service´s "Lov om klage- og erstatningsadgang".

Side effects, risks and disadvantages for patients:

The procedures performed in the project are already performed in detection of COVID-19 infection, and do not involve any known risks of side effects. There may be discomfort associated with the collection of the swab itself, in addition, there is a minor inconvenience for the patients in terms of the time they will have to spend on examination. However, the participants will be citizens who already have booked an appointment for COVID-19 test, and it is therefore expected that they agree with the discomfort or waiting time.

Clinical information from patient records:

Age of the participants, the reason for the booking of appointment at one of Testcenter Denmark's test sites, as well as the results from the PCR test and the rapid antigen test will be registered for all trial participants.

Operating expenses and financial conditions:

No members of the research group behind the project have financial interests in the execution or results of the project. The test staff who are to carry out the swabs for RT-PCT testing are part of Testcenter Danmark's staff and are paid from here. The rapid antigen tests are made available without payment by the distributor (Copenhagen Medical), however they have no role in the design of the project, nor the interpretation of the data.

Application for funding is not planned, but should economical support be obtained anyway, this will be deposited in a foundation account under the Foundation Administration at Rigshospitalet, which is under the hospital's audit.

The Scientific Ethics Committees will be informed and the participant information updated if funding is obtained.

Interruption of the experiment:

The trial will be discontinued in the exceptional circumstances where it is impossible to complete the experiment. Likewise, extraordinary events that render the project incomplete in its entirety will lead to withdrawal for all ongoing trials participants.

Perspectives:

If the sensitivity of the rapid antigen tests is reliable, this may lead to a more widely use of the rapid antigen tests in detection of COVID-19 infection in Denmark. As the response time of the rapid antigen tests is significantly faster than the PCR examinations, it can potentially lead to a faster containment of infection, and thus a better opportunity to bring COVID-19 infection in Denmark under control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Having a scheduled appointment for a COVID-19 test at one of the test centers run by Testcenter Danmark in the Capital Region

Exclusion Criteria:

* Non-fluent in Danish
* Impaired citizen i.e. not capable of an independent self-testing
* Neck breathers (Tracheostomy/laryngectomy patients)
* Nasopharyngeal or oropharyngeal anomalies disallowing sampling using swabs

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3070 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the self-collected rapid antigen test compared to healthcare collected test | 48 hours from sampling to results of RT-PCR analysis
  This applies to both specimen from the anterior part of the nose and from the oropharynx

SECONDARY OUTCOMES:
Diagnostic accuracy including sensitivity and specificity of self-collected and healthcare collected rapid antigen test to RT-PCR tests collected by health care personnel | 30 minutes from sampling to results of the two rapid antigen tests
  These measures apply to both specimen from the anterior part of the nose and from the oropharynx

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine K Jakobsen, MD, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet, Denmark
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet-Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The results will be published as one or more articles in international peer-reviewed scientific papers.

REFERENCES:
- [Background] Jakobsen KK, Jensen JS, Todsen T, Tolsgaard MG, Kirkby N, Lippert F, Vangsted AM, Martel CJ, Klokker M, von Buchwald C. Accuracy and cost description of rapid antigen test compared with reverse transcriptase-polymerase chain reaction for SARS-CoV-2 detection. Dan Med J. 2021 Jun 14;68(7):A03210217. PMID 34169830
- [Background] Bundgaard JS, Raaschou-Pedersen DT, Todsen T, Ringgaard A, Torp-Pedersen C, Von Buchwald C, Iversen K, Bundgaard H. Danish citizens' preferences for at-home oropharyngeal/nasal SARS-CoV-2 specimen collection. Int J Infect Dis. 2021 Aug;109:195-198. doi: 10.1016/j.ijid.2021.06.060. Epub 2021 Jul 1. PMID 34216732
- [Background] McCulloch DJ, Kim AE, Wilcox NC, Logue JK, Greninger AL, Englund JA, Chu HY. Comparison of Unsupervised Home Self-collected Midnasal Swabs With Clinician-Collected Nasopharyngeal Swabs for Detection of SARS-CoV-2 Infection. JAMA Netw Open. 2020 Jul 1;3(7):e2016382. doi: 10.1001/jamanetworkopen.2020.16382. PMID 32697321
- [Background] Lindner AK, Nikolai O, Kausch F, Wintel M, Hommes F, Gertler M, Kruger LJ, Gaeddert M, Tobian F, Lainati F, Koppel L, Seybold J, Corman VM, Drosten C, Hofmann J, Sacks JA, Mockenhaupt FP, Denkinger CM. Head-to-head comparison of SARS-CoV-2 antigen-detecting rapid test with self-collected nasal swab versus professional-collected nasopharyngeal swab. Eur Respir J. 2021 Apr 15;57(4):2003961. doi: 10.1183/13993003.03961-2020. Print 2021 Apr. PMID 33303544
- [Background] Wurstle S, Spinner CD, Voit F, Hoffmann D, Hering S, Weidlich S, Schneider J, Zink A, Treiber M, Iakoubov R, Schmid RM, Protzer U, Erber J. Self-sampling versus health care professional-guided swab collection for SARS-CoV-2 testing. Infection. 2021 Oct;49(5):927-934. doi: 10.1007/s15010-021-01614-9. Epub 2021 May 10. PMID 33970430
- [Background] Tonen-Wolyec S, Dupont R, Awaida N, Batina-Agasa S, Hayette MP, Belec L. Evaluation of the Practicability of Biosynex Antigen Self-Test COVID-19 AG+ for the Detection of SARS-CoV-2 Nucleocapsid Protein from Self-Collected Nasal Mid-Turbinate Secretions in the General Public in France. Diagnostics (Basel). 2021 Nov 27;11(12):2217. doi: 10.3390/diagnostics11122217. PMID 34943454
- [Background] Harmon A, Chang C, Salcedo N, Sena B, Herrera BB, Bosch I, Holberger LE. Validation of an At-Home Direct Antigen Rapid Test for COVID-19. JAMA Netw Open. 2021 Aug 2;4(8):e2126931. doi: 10.1001/jamanetworkopen.2021.26931. PMID 34448871
- [Background] Bundgaard H, Bundgaard JS, Raaschou-Pedersen DET, von Buchwald C, Todsen T, Norsk JB, Pries-Heje MM, Vissing CR, Nielsen PB, Winslow UC, Fogh K, Hasselbalch R, Kristensen JH, Ringgaard A, Porsborg Andersen M, Goecke NB, Trebbien R, Skovgaard K, Benfield T, Ullum H, Torp-Pedersen C, Iversen K. Effectiveness of Adding a Mask Recommendation to Other Public Health Measures to Prevent SARS-CoV-2 Infection in Danish Mask Wearers : A Randomized Controlled Trial. Ann Intern Med. 2021 Mar;174(3):335-343. doi: 10.7326/M20-6817. Epub 2020 Nov 18. PMID 33205991
- [Background] Therchilsen JH, von Buchwald C, Koch A, Dam Nielsen S, Rasmussen DB, Thudium RF, Kirkby NS, Raaschou-Pedersen DET, Bundgaard JS, Iversen K, Bundgaard H, Todsen T. Self-Collected versus Healthcare Worker-Collected Swabs in the Diagnosis of Severe Acute Respiratory Syndrome Coronavirus 2. Diagnostics (Basel). 2020 Sep 9;10(9):678. doi: 10.3390/diagnostics10090678. PMID 32916801
- [Background] Jakobsen KK, Schmidt Jensen J, Todsen T, Lippert F, Cyril ;, Martel J-M, et al. Detection of SARS-CoV-2 infection by rapid antigen test in comparison with RT-PCR in a public setting. medRxiv [Internet]. 2021 Jan 25 [cited 2021 Feb 25];2021.01.22.21250042. Available from: https://doi.org/10.1101/2021.01.22.21250042
- [Derived] Todsen T, Jakobsen KK, Gronlund MP, Callesen RE, Folke F, Larsen H, Ersboll AK, Benfield T, Gredal T, Klokker M, Kirkby N, von Buchwald C. COVID-19 Rapid Antigen Tests With Self-Collected vs Health Care Worker-Collected Nasal and Throat Swab Specimens: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2344295. doi: 10.1001/jamanetworkopen.2023.44295. PMID 38055280
- See also: Analyses of the COVID19 pandemic by Statens Serum Institut — https://covid19.ssi.dk/analyser-og-prognoser/analyser-og-prognoser-for-epidemien-udvikling
- See also: Weekly reports of surveillance data, Denmark — https://covid19.ssi.dk/overvagningsdata/ugentlige-opgorelser-med-overvaagningsdata
- See also: Weekly updates on the COVID19 pandemic by WHO — https://www.who.int/publications/m/item/weekly-operational-update-on-covid-19---21-december-2020
- See also: Collecting Upper Respiratory Specimens for COVID-19 Testing — http://www.urt-sample.com